CLINICAL TRIAL: NCT06371534
Title: A Randomized, Double-blind, Single-dose, Parallel Study to Compare the Pharmacokinetics and Safety of QL2109 and DARZALEX FASPRO® in Healthy Male Adults
Brief Title: A Study Comparing Pharmacokinetic and Safety of QL2109 and DARZALEX FASPRO® in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QL2109-101
Record Dates: First submitted 2024-04-14; First posted 2024-04-17 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-04

CONDITIONS: Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL2109 (Experimental): QL2109, subcutaneous injection 3-5 min D1 (Day 1, single dose)
  Interventions: Drug: QL2109
- DARZALEX FASPRO® (Active Comparator): DARZALEX FASPRO®, subcutaneous injection 3-5 min D1 (Day 1, single dose)
  Interventions: Drug: DARZALEX FASPRO®

INTERVENTIONS:
Drug: QL2109 — subcutaneous injection 3-5 min D1 (Day 1, single dose)
  Arms: QL2109
Drug: DARZALEX FASPRO® — subcutaneous injection 3-5 min D1 (Day 1, single dose)
  Arms: DARZALEX FASPRO®

SUMMARY:
The goal of this clinical trial is to compare the pharmacokinetic and safety similarity of QL2109 with DARZALEX FASPRO® in healthy male volunteers.

Participants will receive a single injection of QL2109/ DARZALEX FASPRO® Researchers will compare pharmacokinetic, safety, and immunogenic similarities between the two groups.

DETAILED DESCRIPTION:
This is a phase I, randomized, double-blind and parallel group clinical trial . The primary objective is to assess the pharmacokinetic similarity of single injections of QL2109 or DARZALEX FASPRO in healthy volunteers.

The secondary objective are to assess the clinical safety and immunogenicity similarity of single injections of QL2109 or DARZALEX FASPRO® in healthy volunteers.

Subjects would receive a single 1800mg#15ml# of QL2109 or DARZALEX FASPRO® injection.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form and fully understand the test content,process and possible adverse reactions, and be able to complete the study according to the test plan requirements;
* Age 18 ~ 50 (inclusive) years , male;
* 65.0 kg≤ body weight ≤90.0 kg and 18.0 kg/m2≤ Body mass index (BMI)

  ≤28.0 kg/m2;
* Agree to use effective contraception throughout the study period (including but not limited to: physical contraception, surgery, abstinence, etc.) until at least 6 months after the study dosing;
* No history of disease or abnormal past medical history is not clinically significant, and the study doctor's judgment has no impact on the trial.

Exclusion Criteria:

* Have been or are currently suffering from any clinically serious disease of the circulatory system, endocrine system, nervous system, digestive system,respiratory system, urogenital system, hematology, immunology, psychiatric and metabolic abnormalities, or any other disease that can interfere with the test results;
* With acute, chronic, or latent infectious diseases within 1 month before administration;
* With known immune system diseases (autoimmune diseases and immunodeficiency diseases), including but not limited to autoimmune hemolytic anemia;
* Has experienced a recent single dermatomal herpes zoster eruption within 6 months before administration;
* Has a history of multi-dermatomal herpes zoster or central nervous system (CNS) herpes zoster during the screening period or before;
* Positive for indirect antiglobulin test (Indirect Coombs test);
* Use of monoclonal antibody, cell therapy, etc. within 6 months before administration, or daratumumab or its analogues or drugs targeting CD38 before administration;
* Use of any medication, including prescription drugs, over-the-counter (OTC) drugs, and Chinese herbal medicines, within 2 weeks before administration;
* History of drug or food allergy, including allergy to any drug or drug excipient used in the study;
* Fear of needles or blood, or difficulty in venous blood collection (history of difficult blood collection or corresponding symptoms and signs, unable to tolerate venipuncture);
* History of blood donation or total blood loss of 200 mL or more within 3 months before administration;
* Participants in clinical trials of any other drug or device within 3 months (or 5 half-lives of the corresponding investigational product if the half-life of the drug is long (5 half-lives > 3 months)) before administration;
* Major surgery within 3 months before signing the ICF;
* Positive for hepatitis B virus antibodies, hepatitis C virus (HCV) antibodies, human immunodeficiency virus (HIV), or treponema pallidum antibodies (Anti-TP);
* History of drug abuse or substance abuse, or positive in urine drug screening;
* Patients who have been vaccinated with attenuated or live virus vaccine (such as Bacille Calmette-Guérin, BCG) or viral vector vaccine within 12 months before the first dose, or who plan to be vaccinated with such vaccines within 12 months after administration;
* Patients who have been vaccinated with vaccines other than the above attenuated or live viral vaccines and viral vector vaccines within 1 month before the first dose, such as inactivated vaccines and recombinant subunit vaccines;
* Subjects with any other conditions that, in the judgment of the investigator, are ineligible for participation in the study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 228 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
AUC0-∞ | 112 day
  To evaluate pharmacokinetic similarity between QL2109 and DARZALEX FASPRO ® after a single subcutaneous injection in healthy volunteers
Cmax | 112 day
  To evaluate pharmacokinetic similarity between QL2109 and DARZALEX FASPRO® after a single subcutaneous injection in healthy volunteers

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China